CLINICAL TRIAL: NCT05695066
Title: Gastric Content After 6 vs 4 Hours of Preoperative Fasting in Children on Enteral Nutrition. A Randomized Controlled Trial Using Gastric Ultrasound
Brief Title: Gastric Content After 6 vs 4 Hours of Preoperative Fasting in Children
Acronym: ENGUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Peter Frykholm, Associate professor, Uppsala University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ENGUS
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Pulmonary Aspiration of Gastric Contents
Keywords: Preoperation fasting; Anaesthesia; Children; Enteral feeding
MeSH Terms: conditions — Respiratory Aspiration of Gastric Contents

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Computerized randomization. Randomization outcome distributed via sealed envelopes. Randomization key stored on secure server.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4H group (Experimental): Patients parents instructed to stop enteral feeding 4 hours before predicted anesthesia induction
  Interventions: Procedure: Preoperative fasting instruction
- 6H group (Active Comparator): Patients parents instructed to stop enteral feeding 6 hours before predicted anesthesia induction
  Interventions: Procedure: Preoperative fasting instruction

INTERVENTIONS:
Procedure: Preoperative fasting instruction — Patients parents instructed to stop enteral feeding at a specified time before predicted anesthesia induction

SUMMARY:
The primary objective of the study is to compare the risk of increased stomach contents after tube feeding (Enteral feeding) 6 and 4 hours before anesthesia using antrum measured by ultrasound.

DETAILED DESCRIPTION:
Children must fast for a certain period of time before anesthesia and surgery to reduce the risk of food residues being vomited up and ending up in the trachea (so-called aspiration). But there are disadvantages to fasting for a long time before an operation, for example the blood sugar level can drop and the body can become dehydrated. Small children risk such side effects to a greater degree than adults, and therefore international work is underway to revise the rules for fasting before surgery.

Enteral feeding children are a special risk group because they are usually completely dependent on tube feeding for nutrition and fluid intake.

ELIGIBILITY:
Inclusion Criteria:

Child on intermittent or continuous enteral nutrition, scheduled for elective procedure requiring general anesthesia

Exclusion Criteria:

Moderate to severe gastrointestinal motility disorder Emergency surgery Anatomical risk factor for pulmonary aspiration such as achalasia or bowel obstruction Parents cannot understand study information due to language barrier

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
CSA | Immediately before anesthesia induction
  Gastric antral surface area

SECONDARY OUTCOMES:
Suctioned GCV | Immediately after intubation
  Gastric content volume suctioned through nasogastric tube after induction

CONTACTS AND LOCATIONS:
Overall Officials: Peter Frykholm, MD PhD, Principal Investigator — Uppsala University Hospital
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Pre-operative fasting in children: A guideline from the European Society of Anaesthesiology and Intensive Care — https://pubmed.ncbi.nlm.nih.gov/34857683/
- See also: Ultrasound assessment of gastric emptying time after a standardised light breakfast in healthy children: A prospective observational study. — https://pubmed.ncbi.nlm.nih.gov/30095551/
- See also: Gastric content assessed with gastric ultrasound in paediatric patients prescribed a light breakfast prior to general anaesthesia: A prospective observational study. — https://pubmed.ncbi.nlm.nih.gov/31608517/